CLINICAL TRIAL: NCT04435561
Title: Efficacy of Dry Needling in the Spasticity of the Hemiparetic Limbs Post-stroke
Brief Title: Efficacy of Dry Needling in the Spasticity Post-stroke
Acronym: DNSpasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMADryNeed
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Spasticity, Muscle
Keywords: dry needling; spasticity; hypertonia; stroke
MeSH Terms: conditions — Muscle Spasticity; Muscle Hypertonia; Stroke | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard physiotherapy rehabilitation and dry needling (Experimental): In addition to the usual therapy, the experimental group will receive the application of dry needling technique in the hemiparetic limbs.
  Dry needling intervention will take place over a period of one and a half months (6 weeks), with a total of 6 sessions. Each session will be performed once a week, where a single puncture will be made in each muscle to be treated, using Hong´s technique and lasting 60 seconds per muscle (or until the muscle is release).
  The muscles that will receive dry needling are the following ones:
  * Upper limb: infraspinatus, teres minor, pectoralis major, deltoid.
  * Lower limb: gastrocnemius, soleus and anterior tibial muscles.
  Interventions: Other: Standard physiotherapy rehabilitation and dry needling
- Standard physiotherapy rehabilitation (Other): The control group will receive the usual therapy and treatment.
  Interventions: Other: Standard physiotherapy rehabilitation

INTERVENTIONS:
Other: Standard physiotherapy rehabilitation and dry needling — The dry needling group receives 6 sessions of dry needling in the spastic muscles of the upper and lower hemiparetic limbs.
  Arms: Standard physiotherapy rehabilitation and dry needling
Other: Standard physiotherapy rehabilitation — This group receives their traditional intervention, without dry needling.
  Arms: Standard physiotherapy rehabilitation

SUMMARY:
Stroke is a serious clinical condition and one of the leading causes of long-term disability in the world. One of the most serious complications of this condition is spasticity. Recently, dry needling has commented to be used as a treatment in muscle spasticity of chronic patients after a stroke, producing improvements in clinical conditions.

This study evaluates the effectiveness of dry needling technique in the spasticity of the hemiparetic limbs in chronic post-stroke patients. The Modified Ashworth Scale is used to measure the spasticity´s improvement after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* First hemiplegic ischemic stroke.
* Chronic stroke (stroke at least 6 months before the trial).
* Present a level of spasticity equal or greater than 1 according to the Modified Asworth Scale.
* Preserve cognitive capacity.
* Being able to understand and follow simple instructions.
* Not afraid of needles.

Exclusion Criteria:

* Recurrent stroke.
* Subjects with cognitive disorders.
* Presenting any medical contraindication for the dry needling procedure or problems with coagulation or epilepsy.
* Alteration of sensitivity.
* Receives nerve block or botulinum toxin treatments in a period equal or less than 6 months, since ir can modify the results.
* Hemorrhagic stroke.
* Subjects who do not consent to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in spasticity | Baseline, 6 weeks of intervention (before and immediately after the treatment) and follow-up 1,3,6 and 12 months after the end of the intervention.
  The spasticity will be measure with the Modified Ashworth Scale. Modified Ashworth Scale is one of the most widely used scales for spasticity measurement. It is an useful, valid and reliable assessment tool that measures the passive movement of a specific joint. It is a valid instrument to represent a quantitative clinical measure of the severity of spasticity in patients with neurological involvement.
  The scale goes from 0 to 4 points. The higher the score, the greater the impact.
  Experimental group: Spasticity will be measure before and immediately after the treatment of dry needling in each session (once a week for 6 weeks) and in a follow-up period after finishing treatment (1,3,6 and 12 months after treatment).
  Control group: Spasticity will be measure at the beginning of the week (before usual therapy) and at the end of the week.

SECONDARY OUTCOMES:
Changes in range of motion | Baseline, 6 weeks of intervention (before and immediately after the treatment) and follow-up 1,3,6 and 12 months after the end of the intervention.
  Active and passive range of motion of the shoulder and ankle will be measure with an standard goniometer. Each movement will be evaluated three times, and the average of theses three results will be performed. The same procedure will be followed to measure both active and passive range of motion of each patient.
  Experimental group: Range of motion will be measure before and immediately after the treatment of dry needling in each session (once a week for 6 weeks) and in a follow-up period after finishing treatment (1,3,6 and 12 months after treatment).
  Control group: Range of motion will be measure at the beginning of the week (before usual therapy) and at the end of the week.
Changes in Motor function of the upper and lower limb | Baseline, 6 weeks of intervention (before and immediately after the treatment) and follow-up 1,3,6 and 12 months after the end of the intervention.
  Fugl-Meyer Scale is one of the most complete quantitative measures designed to measure disability after a stroke. It is divided into five domains and each domain has other elements that are evaluated on an ordinal scale of 0 to 2 points.
  The upper and lower limb motor assessment will be used, with a maximum of 100 points, 66 and 34 respectively, and a minimum of 0 points. The lower the score, the greater the impact.
  Fugl-Meyer Arm Motor Assessment will be use to evaluate motor function of the upper hemiparetic limb and the Fugl-Meyer Motor Leg Assessment to evaluate motor function of the lower hemiparetic limb.
  Experimental group: Motor function will be measure before and immediately after the treatment of dry needling in each session (once a week for 6 weeks) and in a follow-up period after finishing treatment (1,3,6 and 12 months after treatment).
  Control group: Motor function will be measure at the beginning of the week (before usual therapy) and at the end of the week.
Changes in Gait | Baseline, 6 weeks of intervention (before and immediately after the treatment) and follow-up 1,3,6 and 12 months after the end of the intervention.
  The gait will be measure with the Wisconsin Gait Scale. Gait in hemiparetic patients after a stroke must be safe and efficient. Wisconsin Gait Scale is an instrument used to measure gait problems experienced by patients who have hemiplegia after a stroke. This scale can be used as a tool to determine the effectiveness of rehabilitation training and observe how the patient develops in the different phases of gait.
  The maximum score is 42 points and the minimum 13.35 points. The higher the score, the greater the patient´s gait involvement.
  Experimental group: Gait will be measure before and immediately after the treatment of dry needling in each session (once a week for 6 weeks) and in a follow-up period after finishing treatment (1,3,6 and 12 months after treatment).
  Control group: Gait will be measure at the beginning of the week (before usual therapy) and at the end of the week.
Changes in Physical disability | Baseline, 6 weeks of intervention (once a week) and follow-up 1,3,6 and 12 months after the end of the intervention.
  Barthel Index will be used to measure physical disability. It is a widely used instrument to measure the ability of a person to perform daily activities. This tool assesses the independence of the patient to carry out theses activities with or without help. Thanks to this tool, the dependency´s degree can be estimated quantitatively.
  The maximum score is 100 points and the minimum is 0. The higher the score, the more independence the subject will have.
  Experimental group: Physical disability will be measure only before the treatment (is the only one that won´t be measure after each session) of dry needling in each session (once a week for 6 weeks) and in a follow-up period after finishing treatment (1,3,6 and 12 months after treatment).
  Control group: Physical disability will be measure at the beginning of the week (before usual therapy) and at the end of the week.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martin Valero, PhD, Principal Investigator — University of Malaga; Juan Antonio Armenta Peinado, PhD, Study Director — University of Malaga

IPD SHARING:
Plan to Share IPD: No